CLINICAL TRIAL: NCT03658083
Title: Exploring Robotic-assisted Thoracic Surgery for Lung Cancer: Does Robotic-assisted Thoracic Surgery Result in Improved Functional Outcomes Compared to Thoracotomy and How do Patients Appraise the Experience of Undergoing RATS
Brief Title: Exploring Robotic-assisted Thoracic Surgery for Lung Cancer
Acronym: ROSE
Status: Completed | Type: Observational
Sponsor: Teesside University (Other)
Collaborators: South Tees Hospitals NHS Foundation Trust (Other); Barts & The London NHS Trust (Other)
Responsible Party: Principal Investigator, Samantha Harrison, Reader in research, Teesside University
Other Study IDs: 228/16
Record Dates: First submitted 2018-08-29; First posted 2018-09-05 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Lung Cancer; Thoracic Cancer; Surgery
Keywords: exercise; physical activity; quality of life; qualitative; recovery
MeSH Terms: conditions — Lung Neoplasms; Motor Activity | interventions — Thoracotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thoracotomy: Individuals referred for a lung resection via thoracotomy with a primary or secondary diagnosis of lung cancer. Those with a tumor >7cm will be excluded.
  Interventions: Procedure: Thoracotomy
- Robotic-assisted thoracic surgery: Individuals referred for a lung resection via robotic-assisted thoracic surgery with a primary or secondary diagnosis of lung cancer. Those with a tumor >7cm will be excluded.
  Interventions: Procedure: Robotic-assisted thoracic surgery

INTERVENTIONS:
Procedure: Thoracotomy — Open surgery
  Groups: Thoracotomy
Procedure: Robotic-assisted thoracic surgery — Minimally invasive surgery
  Groups: Robotic-assisted thoracic surgery

SUMMARY:
Background Surgery for lung cancer can be performed using open (thoracotomy) or minimally invasive techniques (Video Assisted Thoracic Surgery (VATS)). Despite being associated with fewer postoperative complications (PPCs) VATS is difficult to perform and is only used by 20-44% of thoracic surgeons in the UK. Robotic-Assisted Thoracic Surgery (RATS) maybe a more attractive minimally invasive approach. To date, no studies have explored the impact of RATS on exercise capacity or physical activity and although 1 study has looked at Heath Related Quality of Life (HRQOL) post-RATS compared to an open technique indicators of surgical technique were not controlled for. Furthermore, investigators have little understanding of patients' experience of RATS.

Aims

1. To examine the variability of change in exercise capacity and health-related quality of life (HRQOL) between those who receive thoracotomy V RATS.
2. To compare the difference in post-operative physical activity (step and activity count), across 7 days, in those who receive thoracotomy V RATS.
3. To explore the manner in which patients appraise their experience of undergoing RATS.

Methods:

A mixed-method, multi-center study will be undertaken, utilizing a prospective quasi-experimental study design and an interpretive phenomenological approach. 80 individuals, referred for a lung lobectomy with a primary or secondary diagnosis of lung cancer, will complete outcomes assessed at 4 time-points. The Incremental Shuttle Walk Test (ISWT) and the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30) and the EORTC Lung Cancer module (EORTC QLQ LC13) will be completed at: baseline, 3-6 days post surgery, 6-weeks post-surgery and at 3-month follow up. Patients will wear an activity monitor immediately post-surgery until 1-week post-discharge. Step and activity counts will be recorded. In-depth interviews will be conducted with up to 15 patients who underwent RATS to explore the manner in which patients appraise their experience of RATS.

DETAILED DESCRIPTION:
Lung cancer is the second most common cause of cancer in the UK and the most common cause of cancer death. Surgery is currently the most effective treatment for curing lung cancer and it can be performed using open (thoracotomy) or minimally invasive techniques (Video Assisted Thoracic Surgery (VATS)). Despite VATS being associated with fewer postoperative complications (PPCs), faster recovery and better survival at 4 years compared to thoracotomy it is only used by 20-44% of thoracic surgeons in the UK and just 5% of surgeons in Europe report using minimally invasive techniques for lung resection. Rigid, restrictive instruments and suboptimal vision means a steep learning curve is necessary to conduct VATS successfully. RATS maybe a more attractive minimally invasive approach as it offers 3DHD vision, a 360 degree view of the chest, and a fully articulated arm. JCUH and the Barts Hospital are two of the few centers in the UK performing RATS.

Research on RATS has been largely limited to single retrospective case series reports focusing on safety (PPCs and mortality) and cost effectiveness outcomes. Little research has been conducted exploring the effect of RATS on patient-centered outcomes that are also important quality measures.

To date, no studies have explored the impact of RATS on exercise capacity, yet investigators know that individuals who undergo a thoracotomy have a 16% reduction in exercise capacity at 6 months follow up. Exercise capacity has been shown to be an important predictor for long-term prognosis and length of stay following thoracic surgery, which can have substantial implications for cost. Furthermore, percentage VO2 max has been shown to be the best predictor of PPCs within 30 days of undergoing a lung resection (predictive value 85.5%), which is an important indicator of patient safety.

Two studies have looked at HRQOL post-RATS and compared it to an open technique. Balduyck and colleagues reported that whilst significant reductions from baseline were seen 1 month post-surgery in those who underwent an open procedure (sternotomy), HRQOL had returned to baseline values by 1 month post-surgery in those who underwent RATS. However, indicators of whether individuals received RATS or an open procedure were not controlled for which is likely to be important as individuals who have large tumors are not eligible to receive RATS. Instead RATS is usually assigned to older, frailer individuals. The second study did conduct between-groups comparisons between those who underwent a robotic lobectomy V those who received an open rib and nerve sparing lobectomy. The mental-component of the SF-12 was significantly higher in the robot group at 3 weeks post-surgery, indicating better mental quality of life, although there were no significant between-group differences detected for the physical-component. By 4 months follow up neither the mental nor the physical HRQOL scores differed between the two groups. The SF-12 in a general measure of health status and to date the impact of open surgery V RATS on disease-specific HRQOL has not been explored.

Physical activity is associated with improved HRQOL in patients with lung cancer and increased survival post-diagnosis of cancer. However, 2 months following a lung resection, performed via a thoracotomy or VATS, physical activity levels were still reduced. Unfortunately comparisons between surgical groups were not possible in this study due to the small number of patients who underwent VATS (14), therefore postoperative physical activity in those who have undergone thoracotomy compared to minimally invasive surgery is still unknown.

Clinical Commissioning Group (CCG) outcome indicator set 2015/16 includes enhancing quality of life and ensuring patients have a positive experience of care (NHS England, 2015). To date, no qualitative research exploring the patients' experience of RATS has been conducted and investigators have little understanding of patients' experience of thoracic surgery in general. Interestingly, a very recent study exploring preoperative nurses work experience with robotics found that feelings of uncertainty and concerns about safety were common due to a lack of education about the robot system. It is likely, these feelings of unease are translated to patients during their preoperative consultation leading to heightened anxiety. Furthermore, if nurses do not feel they have sufficient information about the robot system they are unlikely to be educating patients fully about their procedure. A study exploring the appraisals of patients' experience of RATS is important to identify ways in which both pre and postoperative care can be improved.

It would seem literature is scare exploring the impact of RATS on outcomes that are likely to be meaningful to patients. Therefore the overall aim of this study is to examine the impact of RATS compared to thoracotomy on patient-centered outcomes and to explore the individuals' experience of undergoing RATS.

Research strategy

Study design

A mixed-method, multi-center study will be undertaken, utilizing a prospective quasi-experimental study design and an interpretive phenomenological approach.

Inclusion/exclusion criteria

Individuals referred for a lung resection with a primary or secondary diagnosis of lung cancer will be eligible, although those with a tumor >7cm will be excluded. Individuals referred for a lung resection via thoracotomy will be recruited from James Cook University Hospital (JCUH), Middlesbrough and those referred for RATS will be recruited from JCUH or St Bartholomew's hospital, London (Barts).

Recruitment

Once a referral for a lung resection via thoracotomy or RATS is received a cover letter and information sheet, containing details of the study, will be mailed to patients along with their clinic appointment letter. Interested patients will be encouraged to contact a member of the research team, by telephone or email, to discuss the study in more detail. When patients attend their preoperative clinic a member of the clinical team will request permission for a member of the research team to approach them about participation in the study. If individuals would like to participate in the study informed consent will be obtained.

Surgical care

Prior to surgery all patients receive standard physiotherapy consisting of breathing exercises and advice on activities postoperatively.

Three cardiothoracic surgeons, 2 at JCUH and 1 at Barts, will perform lung resections.

Consistent with usual care at JCUH and Barts all individuals will be transferred to sitting at the bedside as soon as possible post-surgery and will be required to walk 150m before being discharged home. At JCUH patients are also required to complete a flight of stairs and cycle for five minutes (with no resistance).

Data collection

Demographic and anthropometric information will be collected at baseline at the preoperative clinic visit including; age, sex, BMI, lung function (forced expiratory volume in one second (FEV1) and forced vital capacity (FVC)), smoking history, comorbidities, cancer stage and grade. Details of the operation (i.e. technique, time, surgeon, post-operative pain management) will be documented. Length of stay, readmissions and PPCs will be recorded at 3 months follow-up. The same criteria will be used to define a PPC as applied by Brocki et al. PPCs will be classified as minor (a score of 1), medium (a score of two) or severe (a score of three). A PPC will be defined as clinically relevant if two or more items are graded as a minor complication (score of 1) or one item is graded as a medium or severe complication (scores ≥2).

Quantitative phase

Outcomes will be assessed at 4 time-points; at baseline in the preoperative clinic (1 day to 2 weeks prior to surgery), day 3 post-surgery, at the follow up postoperative clinic visit (within 6 weeks post-surgery) and at an additional hospital visit which will take place at 3 months. The time taken to complete each assessment will be recorded, we estimate no more than 2 hours will be required to complete the outcome variables (ISWT, the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30) and the EORTC Lung Cancer module (EORTC QLQ LC13)). Individuals will also be requested to wear an activity monitor Actigraph G3TX (Actigraph) immediately post-surgery until 1-week post-discharge. Data will be stored on the cardiothoracic database at JCUH or Barts and on an IBM SPSS statistics database at Teesside University.

Qualitative phase

An interpretive phenomenological approach (IPA) will be applied to the collection and analysis of the qualitative data. IPA aims to understand the lived experience of participants in response to a specific event (i.e. undergoing surgery). Analysis examines in detail how an event is experienced and what meaning is ascribed to that event.

An informal interview schedule consisting of open-ended questions will be developed in conjunction with members of the cardiothoracic team. The questions will be developed to stimulate narratives focusing on the experience of undergoing RATS whilst also permitting other topics, important to the individuals, to be discussed.

In-depth interviews will be conducted on up to 15 patients who underwent RATS. The interviews will be conducted at patient's homes one week following hospital discharge (at the same time the activity monitor is collected). Interviews will be largely patient led, allowing individuals to tell their own story in their own words and at their own pace.

Sample Size and Analysis Plan

Quantitative phase

The primary endpoint is exercise capacity measured by the ISWT (m) completed at patients' 6-week postoperative clinic. Based on the minimal clinically important difference (MCID) (48m) for the ISWT (Singh et al 2008), the between-subjects variability in the measure, and the variability in the change scores (the 7-week reliability). A conventional estimation with 90% power and 2 p=0.05 returned a required sample size of 80 patients, 40 per group. This is based on an ANCOVA analysis model, where invetigators look at the differences in the change in ISWT between groups, adjusted for any imbalance between groups in ISWT performance at baseline

Qualitative phase

Analysis will involve conducting a close line-by-line analysis on each original transcript to explore the claims and understandings of the participants. A second researcher will review the original transcripts before the 'emerging themes' are agreed. Once agreed, 2 researchers will transfer the 'emerging themes' across the entire data set, thereafter referring to them as 'master themes' The final master themes will be presented to a third researcher and agreed. Thematic mapping will be used to develop the relationship between themes. Finally, the findings will be translated into a narrative account with verbatim extracts (quotes) to provide a means of validation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals referred for a lung resection via thoracotomy or RATS with a primary or secondary diagnosis of lung cancer

Exclusion Criteria:

* Tumor >7cm

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Individuals referred for a lung resection with a primary or secondary diagnosis of lung cancer will be eligible, although those with a tumor >7cm will be excluded. Individuals referred for a lung resection via thoracotomy will be recruited from James Cook University Hospital and those referred for RATS will be recruited from James Cook University Hospital or the Barts Health.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Change in exercise capacity assessed using the Incremental Shuttle Walk Test (ISWT) | Baseline to 4-6 weeks post-surgery (visit 2)
  Distance walked in meters

SECONDARY OUTCOMES:
Change in physical activity assessed using an Activity Monitor | Immediately post-surgery to 1-week post-discharge
  Actigraph G3TX. Activity counts will be recorded.
Change in health related quality of life assessed using self-reported questionnaire | Baseline to 3-6 days post-surgery (visit 1)
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30)
Change in disease-specific health related quality of life assess using a self-reported questionnaire | Baseline to 3-6 days post-surgery (visit 1)
  European Organization for Reseach and Treatment of Cancer Quality of Life - Lung Cancer module (EORTC QLQ LC13)
Change in Health related quality of life assessed using self-reported questionnaire | Baseline to 4-6 weeks post-surgery (visit 2)
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30)
Change in disease-specific health related quality of life assessed using self-reported questionnaire | Baseline to 4-6 weeks post-surgery (visit 2)
  European Organization for Reseach and Treatment of Cancer Quality of Life - Lung Cancer module (EORTC QLQ LC13)
Change in health related quality of life assessed using self-reported questionnaire | Baseline to 3 month post-surgery (visit 3)
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30)
Change in disease-specific health related quality of lifeassessed using self-reported questionnaire | Baseline to 3 month post-surgery (visit 3)
  European Organization for Reseach and Treatment of Cancer Quality of Life - Lung Cancer module (EORTC QLQ LC13)
Change in exercise capacity assessed using the Incremental Shuttle Walk Test (ISWT) | Baseline to 3-6days post-surgery (visit 1).
  Distance walked in meters
Change in exercise capacity assessed using the Incremental Shuttle Walk Test (ISWT) | Baseline to 3 months post-surgery (visit 3)
  Distance walked in meters

OTHER OUTCOMES:
Length of hospital stay | 3month follow up
  Days in hospital post-surgery
Hospital readmissions | 3month follow up
  Number of times readmitted to hospital following discharge
Post-operative pulmonary complications | 3month follow up
  Based on criteria applied by Brocki et al. Classified as minor, medium or severe

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Harrison, Principal Investigator — Teesside University
Locations (2):
- United Kingdom (2):
  - Barts Health NHS Trust, London
  - James Cook University Hospital, Middlesbrough

IPD SHARING:
Plan to Share IPD: No